CLINICAL TRIAL: NCT05655494
Title: Precision Clinical Trial Recruitment to Promote Cancer Health Equity Across Florida
Brief Title: A Multilevel Approach to Connecting Underrepresented Populations to Clinical Trials
Status: Recruiting | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB202201399; U01CA274970 (NIH); 24-003323 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2022-10-27; First posted 2022-12-19 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Cancer
Keywords: cancer clinical trial; community health educator; colorectal cancer; breast cancer; lung cancer; prostate cancer; skin cancer; virtual health; mHealth; virtual intervention; gastrointestinal diseases; fibrocystic breast disease; online questionnaire; Spanish-language version; Español; colon cancer
MeSH Terms: conditions — Neoplasms; Colorectal Neoplasms; Breast Neoplasms; Lung Neoplasms; Prostatic Neoplasms; Skin Neoplasms; Gastrointestinal Diseases; Fibrocystic Breast Disease; Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stand-alone Portal: The standard of care condition will include a portal that provides patients with access to existing online cancer clinical trial resources in one location. This includes links to pages with basic information about cancer clinical trials, ongoing studies, enrollment opportunities for existing institutional research registries, and contact information for study coordinators.
  Interventions: Behavioral: Stand-alone Research Portal
- Portal with Virtual Community Health Educator (vCHE): The virtual community health educator condition will provide all information in standard of care with the addition of a virtual community health educator. Patients will have the opportunity to choose which virtual community health educator will provide digital navigation. The choices will include at least four English-speaking and four Spanish-speaking virtual community health educators representing different genders and racial/ethnic backgrounds.
  Interventions: Behavioral: Portal with Virtual Community Health Educator (vCHE)

INTERVENTIONS:
Behavioral: Stand-alone Research Portal — The standard of care condition will include a portal that provides patients with access to existing online cancer clinical trial resources in one location. This includes links to pages with basic information about cancer clinical trials, ongoing studies, enrollment opportunities for existing institutional research registries, and contact information for study coordinators.
  Groups: Stand-alone Portal
Behavioral: Portal with Virtual Community Health Educator (vCHE) — The virtual community health educator condition will provide all information in standard of care with the addition of a virtual community health educator. Patients will have the opportunity to choose which virtual community health educator will provide digital navigation. The choices will include at least four English-speaking and four Spanish-speaking virtual community health educators representing different genders and racial/ethnic backgrounds.
  Groups: Portal with Virtual Community Health Educator (vCHE)

SUMMARY:
The purpose of this study is to pilot test and evaluate an existing tailored ALEX (Agent Leveraging Empathy for eXams) Research Portal to navigate Black and Hispanic adult cancer patients and their family members through referral to cancer clinical trials.

DETAILED DESCRIPTION:
Racial and ethnic minorities represent the fastest growing segment of the United States adult population, yet they remain significantly underrepresented in cancer clinical trials (CCTs). Low trust in clinical research and recruitment approaches that fail to address multilevel barriers to CCT participation are key reasons for minority population underrepresentation. Community health educators (CHEs) improve trust in research among underrepresented populations, yet relying on exclusively on CHE availability can limit intervention reach. Virtual CHEs (vCHEs) improve scalability by extending CHE capabilities and capitalizing on remote recruitment techniques. The purpose of the current project is to increase referral of diverse participants to NCI-supported clinical trials via a culturally responsive, multi-level intervention that utilizes vCHEs to reach diverse populations. The investigators will consolidate existing referral channels within the ALEX Research Portal. ALEX offers a custom experience for clinicians, CHEs, and patients to facilitate CCT referrals. Clinicians can utilize the portal to refer to CCTs; CHEs can use the portal to create an avatar that can provide introductory information to patients and schedule video-conference follow-ups; patients, families, and community members can use the portal to easily navigate to key information and make self-and other-referrals. The ability to streamline information to patients and CCT referrals to study coordinators is expected to improve the overall referral to CCTs. The ALEX Research Portal utilizes the adaptive virtual human technology developed at the University of Florida that provides users with culturally and linguistically tailored CCT information. The ALEX Research Portal will be developed and launched across three distinct geographic areas of Florida (Gainesville, Jacksonville, and Miami). This unique collaborative opportunity will provide access to participants representative of the racial and ethnic diversity of the state as well as cancer centers conducting CCTs associated with national networks [Experimental Therapeutics Clinical Trials Network (ETCTN), National Clinical Trials Network (NCTN)]. Guided by the Interactive Systems Framework for dissemination and implementation, our goal is to increase referrals to CCTs by optimizing the ALEX Research Portal for broad use. The outcome will be an evidence-based intervention that can be widely disseminated to quickly increase the referral of diverse patients to CCTs. This project will be conducted in three phases: (Phase I) establish a baseline of referrals and accrual of diverse participants to CCTs across multiple Florida Center Centers, (Phase 2) adapt and pilot the ALEX Research Portal using a randomized controlled clinical trial, and (Phase 3) scale the intervention by dissemination via the OneFlorida network. The proposed study will result in an empirically-tested vCHE Research Portal for increasing trust in CCTs among diverse populations that can easily be adapted and disseminated across the state to overcome challenges associated with recruiting diverse participants to CCTs.

ELIGIBILITY:
Inclusion Criteria:

* An adult 18 to 100 years of age,
* Able to read English or Spanish at least an eighth-grade level,
* From a racial/ethnic background historically underrepresented in cancer clinical trials (e.g. Blacks or African Americans and/or Hispanics or Latinos),
* Have an email account or the ability to receive texts,
* Willingness to be re-contacted,
* Be a resident of the state of Florida.

Exclusion Criteria:

* Unable to read English or Spanish at least at eighth-grade level
* Does not have an email account or the ability to receive texts
* Unwilling to be re-contacted
* Non resident of the state of Florida.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Black/African American and Latino/Hispanic participants living in Florida.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who self-refer to cancer clinical trials | Within two 2 months of consent
  Patients from underrepresented groups will be recruited in this study and equally randomized into either a) standard-of-care web-based educational portal about clinical trials or a b) a web-based portal that includes a virtual Community Health Educator. Participants in both conditions will have the opportunity to self-refer (operationalized as expressing interest in being contacted) to a cancer clinical trial. The numbers of patients referred to a cancer clinical trial will be collected in both treatment groups and the proportions compared to determine whether adding a virtual Community Health Educator to web-based educational resources about cancer clinical trials will increase referrals of minority patients.
  Patients are assigned into 2 groups, and the outcome measure is the number of self-referrals after treatment divided by the total number of patients for both groups.

SECONDARY OUTCOMES:
Virtual Clinical Health Education (vCHE) preferences | Within two months of consent
  Participants assigned to the portal with the virtual Community Health Educator (vCHE) will be able to choose a vCHE among a set with different characteristics. Data on participant preferences for particular vCHE characteristics will be collected.
  The measure is the count number of the participants that choose the different characteristics of vCHE.
Change in trust in Cancer Clinical Trials | Within two months of consent
  Participants who access the portal will first complete a Clinical Trials Attitudes questionnaire (pre-test) that assesses trust in cancer clinical trials (CCTs). Participants will complete the Clinical Trials Attitudes questionnaire (post-test) after interacting with the vCHE. The Clinical Trials Attitudes questionnaire consists of 14 questions answered on a 5-point scale (strongly agree, agree, neither agree nor disagree, disagree, or strongly disagree)
  The change in responses to the Likert-scale items between the pre-intervention questionnaire and the post-intervention questionnaire will be the change in trust in CCTs.

CONTACTS AND LOCATIONS:
Overall Officials: Janice Krieger, PhD, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - University of Florida, Gainesville, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - University of Miami, Miami, Florida